CLINICAL TRIAL: NCT02021799
Title: The Effect of Nutrition on the Microbiome in Pregnant Women and the Use of Micronutrient Supplemented Probiotic Yogurt to Improve Outcomes
Brief Title: The Effect of Under-nutrition on the Human Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: National Institute for Medical Research, Tanzania (Other Government)
Responsible Party: Principal Investigator, Dr. Gregor Reid, Professor, Western University, Canada
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 102400
Record Dates: First submitted 2013-07-04; First posted 2013-12-27 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Pregnancy
Keywords: Gut microbiome; Vaginal microbiome; Oral microbiome; Human milk microbiome; Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Undernourished Pregnant Women (No Intervention): Pregnant women who are classified as undernourished
- Nourished Pregnant Women (No Intervention): Pregnant women who are classified as healthy
- Overweight/obese Pregnant women (No Intervention): Pregnant women who are classified as obese or overweight
- Undernourished + Yogurt Pregnant Women (Experimental): Pregnant women who are undernourished and selected to receive Moringa and Lactobacillus rhamnosus GR-1 probiotic yogurt. Yogurt contained 4.3 grams of Moringa and 10^8 CFU/mL of Lactobacillus rhamnosus GR-1 as well as Streptococcus thermophilus and Lactobacillus bulgaricus starter cultures.
  Interventions: Dietary Supplement: Moringa and Lactobacillus rhamnosus GR-1
- Nourished + Yogurt Pregnant Women (Experimental): Pregnant women who are healthy and selected to receive Moringa and Lactobacillus rhamnosus GR-1 probiotic yogurt. Yogurt contained 4.3 grams of Moringa and 10^8 CFU/mL of Lactobacillus rhamnosus GR-1 as well as Streptococcus thermophilus and Lactobacillus bulgaricus starter cultures.
  Interventions: Dietary Supplement: Moringa and Lactobacillus rhamnosus GR-1

INTERVENTIONS:
Dietary Supplement: Moringa and Lactobacillus rhamnosus GR-1
  Arms: Nourished + Yogurt Pregnant Women; Undernourished + Yogurt Pregnant Women

SUMMARY:
The purpose of this study is to determine whether a difference exists in the gut, oral, vaginal and human milk microbiome of under-nourished pregnant women as compared to healthy and obese pregnant women. In addition, the investigators are setting out to determine if a micronutrient enriched probiotic yogurt can improve the microbiome and pregnancy outcomes of under-nourished pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 12 weeks pregnant
* between the ages of 18 and 40 years

Exclusion Criteria:

* Less than 12 weeks pregnant

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Characterization of gut, oral, vaginal and human milk microbiomes | Monthly for an average of four months
  Fecal, oral and vaginal samples were collected on a monthly basis for an average of four months. Human milk samples were collected twice; at birth and one week after. Microbial DNA will be extracted with the MoBio PowerSoil 96-well htp kit. Samples will be sequenced and changes determined by 16s rRNA profiling.

SECONDARY OUTCOMES:
Assessment of 48-hour Dietary Recalls | Monthly on average for four months
  Dietary recalls will be assessed for average daily caloric, protein, carbohydrate, fat, calcium, iron, zinc, folate and vitamin intake using ESHA Food Processor SQL software.
Changes in body toxin levels | Before and after intervention (approximately 100 days)
  Body toxin levels (metals, pesticides) by HR-SF-ICP-MS and GC/MS
Changes in blood nutrient levels | before, half-way through and after intervention (approximately 100 days)
  Blood nutrient levels (vitamins, macro and micr-nutrients) will be assessed by HPLC, colorimetric Biuret, chemiluminescence and HR-SF-ICP-MS
Analysis of anthropometric measurements | Monthly on average for four months
  Changes in weight gain, mid-upper arm circumference and hemoglobin levels will be examined and changes will be linked to intervention and non-intervention via statistical analysis.

OTHER OUTCOMES:
Analysis of Anthropometric Measurements | Monthly on Average for 4 months
  Change in the weight gain, mid-upper arm circumference and hemoglobin measurements will be analyzed over the course of study.

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Reid, BSc Hons PhD MBA ARM CCM Dr HS, Principal Investigator — Western University, Canada; Lawson Health Research Institute; Jeremy P Burton, Phd, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Nyerere Dispensary, Buswelu, Tanzania

REFERENCES:
- [Derived] Bisanz JE, Enos MK, Mwanga JR, Changalucha J, Burton JP, Gloor GB, Reid G. Randomized open-label pilot study of the influence of probiotics and the gut microbiome on toxic metal levels in Tanzanian pregnant women and school children. mBio. 2014 Oct 7;5(5):e01580-14. doi: 10.1128/mBio.01580-14. PMID 25293764